CLINICAL TRIAL: NCT06978959
Title: Building Capacity for Youth Mental Wellness: Feasibility and Acceptability for a Mental Health Family Navigator Model for Foster Parents
Brief Title: Family Navigator Plus for Foster Parents
Acronym: FN+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Heather Risser, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00222882
Record Dates: First submitted 2025-05-01; First posted 2025-05-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Intervention
Keywords: foster parents; family navigator; psychoeducation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foster Parents (Experimental): Participants will consist of adult (age 18 and older) foster parents of youth between the ages of 6 and 17 with mental health needs. Participants will be located in Illinois, and be either English or Spanish speaking. Participants will attend a 5-week educational program (one session per week) that aims to support them in understanding child behaviors, finding and access mental health services, communicating with providers, and using technology to find support.
  Interventions: Behavioral: FN+ Intervention

INTERVENTIONS:
Behavioral: FN+ Intervention — Participants will attend 5 one-on-one sessions over the course of 5 weeks; they will meet with a family navigator over video conferencing software (e.g., Zoom). The purpose of each sessions are as follows: 1) Provide an overview of the program and help parents understand their perceptions of child behaviors, 2) Train parents to find, access, and overcome barriers to mental health services, 3) Build parent capacity in understanding how mental health treatment works and how to communicate with providers, 4) Help parents understand the common function of child behaviors, and 5) Train parents to find, evaluate, and use online mental health tools. Participants will complete measures of child symptoms, parent activation, barriers to treatment, and/or satisfaction with the program before the intervention, immediately after the intervention, and 3 months after completing the intervention.

SUMMARY:
The investigators have designed a 5-week Family Navigator Plus (FN+) educational program to support foster parents in better understanding their youth's mental health needs and in finding mental health services. The purpose of this interventional study is to assess the the program's acceptability (e.g., satisfaction, barriers to participation, and burden), utility (e.g., how useful foster parents found the program to be), and feasibility (e.g., number referred who meet eligibility, time to complete assessments, self-reported feasibility). The investigators hypothesize that our program will be acceptable, useful, and feasible for foster parents of youth with mental health needs.

ELIGIBILITY:
Inclusion Criteria:

* Foster parent of a youth between the ages of 6 to 17 with mental health needs
* Parent adopted child from foster care
* Living in Illinois, United States
* English or Spanish speaking
* Has access to internet and videoconferencing

Exclusion Criteria:

- Participated in the FN+ Focus Groups or PROACTIVE Parent Pilot Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | Post-Intervention (Week 5) and 3 Month Follow Up (Week 18)
  The Client Satisfaction Questionnaire (CSQ-8) is an eight-item measure that assesses client satisfaction with services including its quality, utility, and relevance.
Post Session Questionnaire (PsQ) | After Completing Each Session (Weeks 1 - 5)
  The PsQ is a measure we created to assess utility and relevance of session content and materials, and to assess if participants intended to use skills/information learned during that session.

SECONDARY OUTCOMES:
Parent Activation Measure - Mental Health | Baseline (Week 1), Post-Intervention (Week 5), 3 month Follow Up (Week 18)
  The Parent-Patient Activation Measure - Mental Health measures parent activation, defined as the knowledge, ability, and confidence to manage their child's mental health care. It consists of 13 items on a 4-point Likert-type scale ranging from 1-4. Item scores are summed for a total composite score ranging from 13 -52. Composite scores are linearly transformed into scores ranging from 0 - 100. Higher scores indicate higher activation in managing their child's mental health care. PP-PAM-MH internal consistency is adequate, alpha = .89; Item-measures correlations ranged from moderate to large, with a median correlation of .61. The P-PAM-MH is positively correlated with measures of empowerment and negatively correlated with measures of strain.
Barriers to Treatment Participation | Baseline (Week 1), Post-Intervention (Week 5), 3 month Follow Up (Week 18)
  The Barriers to Treatment Participation Scale (BTPS; Kazdin et al., 1997), was designed to assess parent's perceptions of barriers to mental health treatment engagement for their children. The scale consists of two sections. The first section contains four subscales that measure the following constructs: stressors and obstacles that compete with treatment (20 items), treatment demands and issues (10 items), perceived relevance of treatment (8 items), and relationship with the therapist (6 items). Response options for these 44 items range from 1 (Never a problem) to 5 (Very often a problem). The second section includes 14 discrete events associated with early treatment termination. Response options for this section include yes and no. Higher scores on the measure indicate more barriers to treatment participation. Scores on the BTPS have been associated with multiple indices measuring the child's participation in treatment. Internal consistency for total score is α =.95, and subscales r
PROMIS-Parent Proxy Pediatric Depressive Symptoms Short Form 8a (parent-report) | Baseline (Week 1), Post-Intervention (Week 5), 3 month Follow Up (Week 18)
  The PROMIS Parent Proxy Depressive Symptoms Short Form 8a measures negative mood and views of self, social cognition, and decreased positive affect and engagement in pediatric populations aged 5- to 17-years old (Irwin, et al., 2012). Parents respond to 8 items assessing their child's symptoms of depression. Response options range from 1 (never) to 5 (almost always). Higher scores indicate higher levels of depressive symptoms. Scores are reported as T-scores ranging from 35-82, with a mean of 50 and standard deviation of 10 in the sample referenced (Irwin et al, 2010). Higher scores indicate higher levels of depressive symptoms. Parent proxy measures were created using Item Response Theory to support theoretically maximized reliability and validity across the trait being measured. Parent proxy scores were strongly univocal with 89% of the general variance explained by the scale's general factor. Internal consistency is adequate at .90.
PROMIS-Parent Proxy Pediatric Anxiety Short Form 8a (parent-report) | Baseline (Week 1), Post-Intervention (Week 5), 3 month Follow Up (Week 18)
  The PROMIS Parent Proxy Anxiety Short Form 8a measures symptoms of fear, anxious misery, hyperarousal, and somatic symptoms related to arousal among pediatric populations aged 5- to 17-years old (Irwin, et al., 2012). Parents respond to 8 items assessing their child's symptoms of anxiety. Response options range from 1 (never) to 5 (almost always). Higher scores indicate higher levels of anxiety. Scores are reported as T-scores ranging from 32-84, with a mean of 50 and standard deviation of 10 in the sample referenced (Irwin et al, 2010). Higher scores indicate higher levels of anxiety. The measure was created using Item Response Theory to support theoretically maximized reliability and validity across the trait being measured. The parent proxy version was validated against other proxy measures to ensure content and discriminant validity. Parent proxy scores were strongly univocal with 87% of the general variance explained by the scale's general factor. Internal consistency = .90.
Pediatric Symptoms Checklist - 17 (Parent Report) | Baseline (Week 1), Post-Intervention (Week 5), 3 month Follow Up (Week 18)
  The Pediatric Symptom Checklist - 17 (PSC-17) was designed to assess psychosocial function in children. The measures includes three subscales that assess symptoms associated with internalizing, externalizing, and attention problems. Response options range from 0 (Never) to 2 (Often). The parent report version is used with children aged 5- to 17- years. T scores range from 0-34, with at or above 15 indicating the presence of a psychosocial impairment. Internalizing or Attention subscale scores at or above 5, and Externalizing scores at or above 7, indicate impairment. The measure has been validated in the general child population. Parent-reported internal consistency range from .79-.83, and overall reliability as .89. A large-scale replication study confirmed reliability was high, with both internal consistency and test-retest reliability both at, or above, 0.85 on the parent report form.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Risser, PhD, Principal Investigator — Northwestern University; Enrollment Contact, If interested in participation, Study Director — Northwestern University email FNplus@northwestern.edu
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NIMH Data Sharing policy, de-identified IDP will be shared in the NIMH Data Archive (NDA, https://nda.nih.gov/)
Time Frame: Per NIMH Data Sharing policy
Access Criteria: Per NIMH Data Sharing policy
URL: https://nda.nih.gov

REFERENCES:
- [Background] Risser, H. J., Morford, A. E., Murphy, A. N., Pinkerton, L. M., Law, C., Yang, Y., ... & Boisseau, C. L. (2024). Feasibility and acceptability of a family navigator program to support foster parents of youth with mental health concerns. Children and Youth Services Review, 160, 107578.